CLINICAL TRIAL: NCT02382575
Title: Efficacy and Safety of Rituximab to That of Calcineurin Inhibitors in Children With Steroid Resistant Nephrotic Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nilratan Sircar Medical College (Other Government)
Responsible Party: Principal Investigator, Dr. Biswanath Basu, Assistant Professor & In charge, Division of Pediatric Nephrology, Nilratan Sircar Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PednephroRCT/PM/NRSMCH-33; CTRI/2015/01/005364 (Registry Identifier: Clinical Trial Registry of India)
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab; Tacrolimus; Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Active Comparator): Tacrolimus: Standard dose with oral Tacrolimus 0.2 mg/kg/day in two divided doses till 6 month of relapse free survival.
  Interventions: Drug: Tacrolimus
- Rituximab (Experimental): Two to four rituximab infusions (over 2-4 weeks) will be administered once every week at standard dose (Intravenous infusion of rituximab 375mg/mt2)depending on circulating B cells level.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Two to four rituximab infusions (over 2-4 weeks) will be administered once every week at standard dose (Intravenous infusion of rituximab 375mg/mt2)depending on circulating B cells level.
  Other Names: anti CD20 monclonal antibody
  Arms: Rituximab
Drug: Tacrolimus — Standard dose with oral Tacrolimus 0.2 mg/kg/day in two divided doses till 6 month of relapse free survival.
  Other Names: Calcineurin inhibitor
  Arms: Tacrolimus

SUMMARY:
The vast majority of children with idiopathic nephrotic syndrome respond well to corticosteroid treatment. However, as many as 20% experience a more complicated course with steroid resistance (SRNS). Repeated and prolonged courses of steroids in these children often result in long-term complications. The goal of treatment is to reduce the rate of relapses, the cumulative dose of corticosteroids, and the incidence of serious complications. In order to minimize the side effects of steroid therapy, different steroid sparing agents such as cyclophosphamide, calcineurin inhibitors(CNI), levamisole, and mycophenolate mofetil (MMF) have been used in SRNS. Whereas CNI are usually considered the steroid sparing drug class of first choice, rituximab is increasingly used as alternative to minimize CNI toxicity. Various prospective studies suggest that Rituximab, a B cell depleting monoclonal antibody, could be a safe and effective alternative to steroid or immunosuppressants to achieve and maintain remission in this population. Rituximab infusion have been shown to be efficacious for 6 to 12 months and the side effect profile observed to date is very benign. Studies comparing the usefulness of these agents are lacking. In this proposed randomized controlled trial, the investigators want to compare the efficacy and safety of CNI to that of Rituximab in treating children with SRNS.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 16 years with SRNS
* Minimal Change disease/Messengioproliferative glomerulonephritis/Focal segmental glomerulosclerosis as per Kidney Biopsy report.
* Estimated glomerular filtration rate (eGFR) >80 ml/min per 1.73 m2 at study entry.
* Not received any steroid sparing agent previously.
* Parents willing to give informed written consent.
* Ability to swallow tablet

Exclusion Criteria:

* Known etiology (e.g., lupus erythematosus, IgA nephropathy, amyloidosis, malignancy, other secondary forms of NS)
* Patients with severe leucopenia (leucocytes <3.0× 1000 cells/mm3), severe anemia (haemoglobin <8.9 g/dl), thrombocytopenia (platelet <100.0 × 1000 cells/mm3) or deranged liver function tests (AST or ALT to >50 IU/L ) at enrolment.
* Known active chronic infection (tuberculosis, HIV, hepatitis B or C)
* Live vaccination within 1 mo

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2015-03-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
12-month relapse-free survival in the intention-to-treat population | 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Biswanath Basu, Principal Investigator — Assistant Professor
Locations (1):
- NRS Medical College & Hospital, Kolkata, West Bengal, India

REFERENCES:
- [Derived] Liu ID, Willis NS, Craig JC, Hodson EM. Interventions for idiopathic steroid-resistant nephrotic syndrome in children. Cochrane Database Syst Rev. 2025 May 8;5(5):CD003594. doi: 10.1002/14651858.CD003594.pub7. PMID 40337980